CLINICAL TRIAL: NCT03078010
Title: Rational Use of Broad-spectrum Antibiotics as Empiric Antibiotic Therapy in Febrile Neutropenia in Recipients of Allogeneic Hematopoietic Cell Transplantation
Brief Title: Choosing the Best Antibiotic to Protect Friendly Gut Bacteria During the Course of Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-097
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Intestinal Microbiome; Febrile Neutropenia
Keywords: Antibiotic; piperacillin-tazobactam; cefepime; aztreonam; 17-097
MeSH Terms: conditions — Febrile Neutropenia | interventions — Piperacillin, Tazobactam Drug Combination; Cefepime

STUDY DESIGN:
Intervention Model Description: This is a randomized open-label phase II study to assess the association between antibiotic treatment strategies and the change in the relative abundance of Clostridiales.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Piperacillin-tazobactam (Active Comparator)
  Interventions: Drug: Piperacillin-tazobactam
- cefepime (Experimental)
  Interventions: Drug: cefepime

INTERVENTIONS:
Drug: Piperacillin-tazobactam — piperacillin-tazobactam (4.5 gm IV q 6 hrs)
  Arms: Piperacillin-tazobactam
Drug: cefepime — (2 gm IV q 8 hrs)
  Arms: cefepime

SUMMARY:
The purpose of this study is to see how different antibiotics affect the community of friendly bacteria existing in the intestinal tract (gut). Under normal circumstances, these friendly bacteria are not harmful and they help with normal bodily functions such as digestion. When these bacteria are absent, several complications may occur, such as infections with harmful bacteria or other inflammatory reactions, that can complicate the stem cell transplant course. Treatment with antibiotics or chemotherapy is known to kill off these friendly bacteria. In this study we compare the effects of different antibiotics on the community of friendly bacteria in the gut. For microbiota-related biomarker analysis, optional urine samples (MSKCC patients only) will be collected at baseline, 7 +/-2 days after initiation of antibiotic therapy, and on post-transplant days +28, +56 and +100 (+/- 7days).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with any hematologic malignancy undergoing

Exclusion Criteria:

* Patients with severe allergies to piperacillin-tazobactam, cefepime, aztreonam or vancomycin. Severe reactions include anaphylaxis and Stevens-Johnson syndrome (SJS)/toxic epidermal necrolysis (TEN).
* Patients with unconfirmed allergies to piperacillin-tazobactam, cefepime, aztreonam or vancomycin can be evaluated by an Allergy/Immunology specialist, after which they may become eligible by a consensus of the treating physician, trial investigator and and the Allery
* Prolonged antibiotic treatment ( ≥10 days, within 3 weeks of enrollment) as prevention or suppression of an ongoing infection, where treatment involves gut-perturbing anti anaerobic antibiotics
* Patients with history of infection with extended-spectrum beta-lactamase producing organism. Patients known to be colonized with multi-drug resistant gram-negative organisms or with history of infection with multi-drug resistant organisms will be evaluated case by case and discussed with infectious disease specialist before enrollment
* Febrile patients
* Patients with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
measurement of fold-change in Clostridiales abundance | 7 +/- 2 days after initiation of piperacillin-tazobactam or cefepime
  Fold change will be assessed 7 +/- 2 days after initiating antibiotic treatment for febrile neutropenia and will be compared to the pre-treatment specimen. Pre-treatment stool specimen will be collected between the time of enrollment Patients will be enrolled and infusion of allografts or first episode of neutropenic fever, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Seo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm